CLINICAL TRIAL: NCT04009096
Title: A Phase IIa Challenge Study to Assess Efficacy of the Plasmodium Vivax Malaria Vaccine Candidates ChAd63 PvDBP and MVA PvDBP in Healthy Adults Living in the UK
Brief Title: VAC071: A Study to Assess Efficacy of the ChAd63/MVA PvDBP Vaccines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC071
Record Dates: First submitted 2019-07-03; First posted 2019-07-05 (Actual); Results first posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2022-09

CONDITIONS: Malaria, Vivax
Keywords: PvDBP; efficacy
MeSH Terms: conditions — Malaria, Vivax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): 3 volunteers receiving 5 x 10^10 vp ChAd63 PvDBP and 2 x 10^8 pfu MVA PvDBP 8 weeks later, in a heterologous prime-boost regimen, followed by blood-stage CHMI 2-4 weeks later.
  Interventions: Biological: ChAd63 PvDBP and MVA PvDBP
- Group 2 (Experimental): Up to 10 volunteers receiving one dose of 5 x 10^10 vp ChAd63 PvDBP, 12-18 months later receiving a second dose of 5 x 10^10 vp ChAd63 PvDBP and 8 weeks later 2 x 10^8 pfu MVA PvDBP, followed by blood-stage CHMI 2-4 weeks later.
  Interventions: Biological: ChAd63 PvDBP and MVA PvDBP
- Group 3 (Experimental): If fewer than 6 volunteers complete the study in Group 2, then new volunteers will be recruited into Group 3, to make up a total of 6 volunteers between Groups 2 and 3 who complete all vaccinations and CHMI.
  Volunteers in Group 3 will receive 5 x 10^10 vp ChAd63 PvDBP and 2 x10^8 pfu MVA PvDBP 8 weeks later, in a heterologous prime-boost regimen, followed by blood-stage CHMI 2-4 weeks later.
  Interventions: Biological: ChAd63 PvDBP and MVA PvDBP

INTERVENTIONS:
Biological: ChAd63 PvDBP and MVA PvDBP — one dose of 5 x 10^10 vp ChAd63 PvDBP and one dose of 2 x 10^8 pfu MVA PvDBP 8 weeks later, in a heterologous prime-boost regimen.

SUMMARY:
This is an open label, Phase IIa, controlled human malaria infection (CHMI) study aimed to assess whether the new vivax malaria vaccines ChAd63 PvDBP and MVA PvDBP can protect against malaria infection.

The participants will receive one or two doses of ChAd63 PvDBP followed by one dose of MVA PvDBP 8 weeks later.

Approximately 4 weeks after the second vacccination, the volunteers will be challenged (deliberately infected) with malaria by intravenous injection blood-stage

DETAILED DESCRIPTION:
Volunteers will be recruited and vaccinated at the CCVTM, Oxford.

There will be two groups vaccinated in the trial, with an optional third group included if fewer than 6 volunteers complete group 2. Up to 19 volunteers will be included in total. These will be compared to a matched number of infectivity controls, receiving no vaccination, who will be recruited as part of a separate study (VAC069 - NCT03797989).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18 to 45 years.
* Red blood cells positive for the Duffy antigen/chemokine receptor (DARC).
* Normal serum levels of Glucose-6-phosphate dehydrogenase (G6PD).
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Willing to allow the Investigators to discuss the volunteer's medical history with their General Practitioner.
* Women only: Must practice continuous effective contraception* for the duration of the study
* Agreement to permanently refrain from blood donation
* Written informed consent to participate in the trial.
* Reachable (24/7) by mobile phone during the period between CHMI and completion of all antimalarial treatment.
* Willing to take a curative anti-malarial regimen following CHMI.
* Willing to reside in Oxford for the duration of the study, until antimalarials have been completed.
* Answer all questions on the informed consent quiz correctly.

  * Female volunteers are required to use an effective form of contraception during the course of the study as malaria challenge could pose a serious risk to both maternal health and the unborn foetus.

Exclusion Criteria:

* History of clinical malaria (any species).
* Travel to a clearly malaria endemic locality during the study period or within the preceding six months.
* Current or planned treatment with long-acting immune-modifying drugs at any time during the study period (e.g. infliximab).
* Chronic use of antibiotics with antimalarial effects (e.g. tetracyclines for dermatologic patients, trimethoprim-sulfamethoxazole for recurrent urinary tract infections, etc.).
* Weight less than 50kg, as measured at the screening visit.
* Receipt of immunoglobulins within the three months prior to planned administration of the vaccine candidate.
* Receipt of blood products (e.g., blood transfusion) at any time in the past.
* Peripheral venous access unlikely to allow twice daily blood testing (as determined by the Investigator).
* Receipt of an investigational product in the 30 days preceding enrolment, or planned receipt during the study period.
* Receipt of any vaccine in the 30 days preceding enrolment, or planned receipt of any other vaccine within 30 days preceding or following each study vaccination, with the exception of licensed COVID-19 vaccines, which should not be received within 14 days before or 7 days after any study vaccination.
* Planned receipt of a COVID-19 vaccine between 2 weeks before the day of CHMI until completion of antimalarial treatment
* Concurrent involvement in another clinical trial or planned involvement during the study period.
* Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data or the P. vivax parasite as assessed by the Investigator.
* History of sickle cell anaemia, sickle cell trait, thalassaemia or thalassaemia trait or any haematological condition that could affect susceptibility to malaria infection.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine e.g. egg products, Kathon, aminoglycosides.
* History of allergic disease or reactions likely to be exacerbated by malaria infection.
* History of clinically significant contact dermatitis.
* Any history of anaphylaxis in reaction to vaccinations.
* Pregnancy, lactation or intention to become pregnant during the study.
* Use of medications known to cause prolongation of the QT interval and existing contraindication to the use of Malarone.
* Use of medications known to have a potentially clinically significant interaction with Riamet and Malarone.
* Any clinical condition known to prolong the QT interval.
* History of cardiac arrhythmia, including clinically relevant bradycardia.
* Disturbances of electrolyte balance, e.g. hypokalaemia or hypomagnesaemia.
* Family history of congenital QT prolongation or sudden death.
* Contraindications to the use of both of the proposed anti-malarial medications; Riamet Malarone.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition that may affect participation in the study.
* Any other serious chronic illness requiring hospital specialist supervision.
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 25 standard UK units every week.
* Suspected or known injecting drug abuse in the 5 years preceding enrolment.
* Hepatitis B surface antigen (HBsAg) detected in serum.
* Seropositive for hepatitis C virus (antibodies to HCV) at screening or (unless has taken part in a prior hepatitis C vaccine study with confirmed negative HCV antibodies prior to participation in that study, and negative HCV RNA PCR at screening for this study).
* Positive family history in both 1st AND 2nd degree relatives < 50 years old for cardiac disease.
* Volunteers unable to be closely followed for social, geographic or psychological reasons.
* Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination. In the event of abnormal test results, confirmatory repeat tests will be requested. Procedures for identifying laboratory values meeting exclusion criteria are shown in SOP VC027.
* Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.
* Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Minassian, MBBS MA DPhil MRCP FRCPath, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology & Tropical Medicine, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Hou MM, Barrett JR, Themistocleous Y, Rawlinson TA, Diouf A, Martinez FJ, Nielsen CM, Lias AM, King LDW, Edwards NJ, Greenwood NM, Kingham L, Poulton ID, Khozoee B, Goh C, Mac Lochlainn DJ, Salkeld J, Guilotte-Blisnick M, Huon C, Mohring F, Reimer JM, Chauhan VS, Mukherjee P, Biswas S, Taylor IJ, Lawrie AM, Cho JS, Nugent FL, Long CA, Moon RW, Miura K, Silk SE, Chitnis CE, Minassian AM, Draper SJ. Impact of a blood-stage vaccine on Plasmodium vivax malaria. medRxiv [Preprint]. 2022 May 30:2022.05.27.22275375. doi: 10.1101/2022.05.27.22275375. PMID 35664997

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3
Started | 3 | 10 | 3
Completed | 3 | 2 | 3
Not Completed | 0 | 8 | 0
Not completed — Withdrawal by Subject | 0 | 7 | 0
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 3 | 10 | 3 | 16
Age, Continuous [Mean (Full Range); unit: years] | 32 [29 to 38] | 28 [20 to 44] | 25 [21 to 29] | 28 [20 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 1 | 7
  Male | 1 | 6 | 2 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 7 | 3 | 13
  Arab | 0 | 1 | 0 | 1
  Asian | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 3 | 10 | 3 | 16

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of the ChAd63 and MVA PvDBP Vaccines, Administered in a Heterologous Prime-boost Regimen, Assessed by a Reduced Parasite Multiplication Rate in Vaccinated Subjects
Description: Quantitative PCR-derived parasite multiplication rate (PMR) will be the primary efficacy endpoint and a comparison of the endpoint between Groups 1, 2 and 3 (pooled data) and malaria-naïve controls partaking in simultaneous CHMI, under identical conditions, will constitute the primary analysis for efficacy.
Time Frame: 3 months post CHMI
Population: Primary efficacy analysis conducted as per protocol on pooled data from all volunteers across groups 1, 2 and 3 who underwent CHMI. Numbers in each group too small for meaningful summary statistics to be reported for each group separately.
Measure: Median (Full Range); unit: parasite multiplication rate per 48hr
Groups:
- Groups 1, 2 and 3 Volunteers Completing CHMI: Pooled data of all volunteers in Groups 1, 2 and 3 who underwent CHMI
Arm/Group | Groups 1, 2 and 3 Volunteers Completing CHMI
Number analyzed (Participants) | 8
parasite multiplication rate per 48hr | 5.4 [4.0 to 7.3]
Statistical Analysis 1: Comparison: Groups 1, 2 and 3 Volunteers Completing CHMI; Comparison of pooled data from Groups 1, 2 and 3 volunteers who completed CHMI with pooled data of infectivity controls (unvaccinated) from CHMI study running in parallel (VAC069 study); Test type: Other; p = 0.14, Wilcoxon (Mann-Whitney) — Two tailed p value reported for Mann-Whitney test comparing controls with each vaccinees

2. Secondary Outcome: Safety of the ChAd63 and MVA PvDBP Vaccines Andidates, Administered in a Heterologous Prime-boost Regimen in a CHMI Study in Healthy Volunteers
Description: No of participants reporting adverse event
Time Frame: Within 28 days following each vaccination. Vaccinations occurred at 0 and 2 months in Groups 1 and 3 (ChAd63, MVA PvDBP); and at 0, 17 and 19 months in Group 2 (ChAd63, ChAd63, MVA PvDBP).
Population: Adverse events following vaccinations are analysed by IMP administered
Measure: Count of Participants; unit: Participants
Groups:
- Following ChAd63 PvDBP Vaccination: Volunteers who received at least one dose of ChAd63 PvDBP
- Following MVA PvDBP Vaccination: Volunteers who received vaccination with MVA PvDBP
Arm/Group | Following ChAd63 PvDBP Vaccination | Following MVA PvDBP Vaccination
Number analyzed (Participants) | 16 | 8
Participants
  Any grade 3 solicited adverse event | 1 | 2
  Any grade 3 unsolicited adverse event | 0 | 0
  Any grade 3 laboratory adverse event | 1 | 0

3. Secondary Outcome: The Humoral Immunogenicity ChAd63 and MVA PvDBP Vaccine Candidates, Administered in a Heterologous Prime-boost Regimen
Description: Total IgG antibody response to the P. vivax Duffy-binding protein (PvDBP)
Time Frame: 14 days after the final vaccination. Final vaccinations (MVA PvDBP) occurred at 2 months in Groups 1 and 3; and at 19 months in Group 2.
Population: Immunological analysis conducted as per protocol on pooled data from all volunteers across groups 1, 2 and 3 who completed vaccinations. Numbers in each group too small for meaningful summary statistics to be reported for each group separately.
Measure: Geometric Mean (Full Range); unit: μg/mL
Groups:
- Groups 1, 2 and 3 Volunteers: Pooled data of all volunteers in Groups 1, 2 and 3 who completed vaccinations
Arm/Group | Groups 1, 2 and 3 Volunteers
Number analyzed (Participants) | 8
μg/mL | 29 [9 to 85]

4. Secondary Outcome: The Cellular Immunogenicity ChAd63 and MVA PvDBP Vaccine Candidates, Administered in a Heterologous Prime-boost Regimen
Description: PvDBPII-specific CD4+ CD45RA- CCR7- effector memory T cells producing IFN-γ
Time Frame: 14 days after the final vaccination. Final vaccinations (MVA PvDBP) occurred at 2 months in Groups 1 and 3 ; and at 19 months in Group 2.
Population: as for outcome 3
Measure: Mean (Full Range); unit: Percentage of IFN-γ+ cells
Arm/Group | Groups 1, 2 and 3 Volunteers
Number analyzed (Participants) | 8
Percentage of IFN-γ+ cells | 0.6825 [0.09500 to 1.951]

5. Secondary Outcome: Immunological Readouts for Association With a Reduced Parasite Multiplication Rate
Description: Statistical correlation between anti-PvDBP antibody responses induced by the ChAd63 and MVA PvDBP vaccines and PMR.
Time Frame: 3 months post CHMI
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Data on solicited adverse events were collected for 7 days after vaccination and unsolicited adverse events for 28 days post-vaccination. Serious adverse events were collected for the study duration: up to 12 months for Group 1 and 3 participants, and up to 29 months for Group 2 participants.
Description: Following each vaccination, volunteers completed an electronic diary card for 28 days with adverse event data. Solicited AEs, collected for 7 days, included local AEs (pain, erythema, warmth, swelling and itching) and systemic AEs (headache, malaise, myalgia, arthralgia, feverishness, nausea, fatigue, and measured fever
Arm/Group | Following ChAd63 PvDBP Vaccination | Following MVA PvDBP Vaccination
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/8
Other Adverse Events (participants affected / at risk) | 2/16 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Following ChAd63 PvDBP Vaccination (N=16) | Following MVA PvDBP Vaccination (N=8)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 0
Feverish (General disorders) | 0 | 1
Fever (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/96/NCT04009096/Prot_SAP_000.pdf